CLINICAL TRIAL: NCT01591590
Title: Correlating the Tumoral Metabolic Progression Index Measured by Serial FDG PET-CT and Apparent Diffusion Coefficient Measured by MRI to Patient's Outcome in Advanced Colorectal Cancer
Brief Title: Correlating the Tumoral Metabolic Progression Index to Patient's Outcome in Advanced Colorectal Cancer
Acronym: CORIOLAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CORIOLAN; 2011-006280-21 (EudraCT Number)
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Cancer; Colon Cancer; Rectal Cancer; PET; PET-CT; MRI; Diffusion MRI; Apparent Diffusion Coefficient; ADC; Metabolic Progression Index
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Diffusion Tensor Imaging; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Experimental): This is an Interventional, Non Therapeutic arm
  Interventions: Other: FDG PET-CT; Other: Diffusion MRI; Other: Blood samples (plasma preparation and CTC)

INTERVENTIONS:
Other: FDG PET-CT — All patients will undergo FDG PET-CT at inclusion and 2 weeks after
  Other Names: Metabolic Investigation
Other: Diffusion MRI — All patients will undergo Diffusion MRI at inclusion and 2 weeks later
  Other Names: Metabolic Investigation
Other: Blood samples (plasma preparation and CTC)

SUMMARY:
The purpose of this study is to assess whether in a population of patients with advanced colorectal cancer for which no known effective therapy is available, measuring the spontaneous evolution of tumoral metabolic progression index by serial FGD PET-CT and Diffusion MRI can show that tumor growth rate is related to the patient's outcome, and that serial FDG PET-CT and Diffusion MRI are able to measure it.

DETAILED DESCRIPTION:
Natural history of tumors is a poorly studied subject, the clinical evidence of some tumors aggressiveness as opposed to some other's indolent behavior has never been formally assessed in daily practice or in clinical studies and remains largely unpredictable. The patient's populations are in fact a mix between different tumoral phenotypes that while carrying the same apparent disease evolve with different outcomes.

We hypothesize that,in a population of patients with advanced colorectal cancer for which no known effective therapy is available, measuring the spontaneous evolution of tumoral metabolic progression index by serial FGD PET-CT and Diffusion MRI can show that tumor growth rate is related to the patient's outcome, and that serial FDG PET-CT and Diffusion MRI are able to measure it.

If the hypothesis is verified, this finding could:

* Allow to define therapeutic strategies according to the tumoral metabolic progression index.
* Limit the need for randomization in the early drug development phases as each patient could be considered as his own control.
* To stratify patients according to their baseline metabolic growth rate in randomized controlled trials with overall survival as an endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed colorectal cancer that is metastatic or unresectable and for which standard treatments do not exist or are no longer effective.
* The tumor should be refractory to all standard chemotherapy agents (fluoropyrimidines, irinotecan, and oxaliplatin) and anti-EGFR monoclonal antibodies in case of wild type Kras (cetuximab or panitumumab) administered before study entry. Prior treatment with bevacizumab, regorafenib and/or aflibercept is allowed but not mandatory
* Participants should be candidate for a Phase I study
* Age equal or over 18 years.
* Life expectancy of greater than 12 weeks.
* ECOG performance status ≤ 1.
* Participants must have normal organ and marrow function as defined below:

Total bilirubin within 2 × normal institutional upper limits AST/ALT/Alk Phosphatase levels < 5 × normal institutional upper limits Creatinine within 2 × normal institutional upper limits or creatinine clearance > 35mL/min

* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry during the assessment. For women of childbearing potential a pregnancy test (urinary or serum) must be performed within 7 days prior to inclusion and it must be negative. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately within one month.
* Signed written informed consent obtained prior to any study specific screening procedures).

Exclusion Criteria:

Patients who exhibit any of the following conditions at screening will not be eligible for admission into the study:

* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Participants who have had a major surgery or radiotherapy within 4 weeks prior to entering the study.
* Patients receiving any experimental agents during the assessment time period.
* Patients with uncontrolled brain metastases.
* Bleeding diathesis, history of cardiovascular ischemic disease or cerebrovascular incident within the last six months.
* Participants who have had a major surgery or radiotherapy within 4 weeks prior to entering the study
* Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness or any significant disease which, in the investigator's opinion, would exclude the patient from the study.
* Pregnancy or breastfeeding before the FDG PET-CT scan examinations
* Uncontrolled Diabetes.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Contra-indications to the use of MRI: cardiac stimulator, implanted cardiac wires, any implanted electronic devices, intra-ocular metallic foreign bodies.
* Medical, geographical, sociological, psychological or legal conditions that would not permit the patient to complete the study or sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-06; Primary Completion 2019-07 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months

SECONDARY OUTCOMES:
Tumour Progression | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amélie Deleporte, MD, Principal Investigator — Jules Bordet Institute , Universite Libre De Bruxelles
Locations (1):
- Jules Bordet Institute, Brussels, Belgium

REFERENCES:
- [Derived] Deleporte A, Paesmans M, Garcia C, Vandeputte C, Lemort M, Engelholm JL, Hoerner F, Aftimos P, Awada A, Charette N, Machiels G, Piccart M, Flamen P, Hendlisz A. Correlating tumor metabolic progression index measured by serial FDG PET-CT, apparent diffusion coefficient measured by magnetic resonance imaging (MRI) and blood genomics to patient's outcome in advanced colorectal cancer: the CORIOLAN study. BMC Cancer. 2014 May 30;14:385. doi: 10.1186/1471-2407-14-385. PMID 24885112
- See also: Jules Bordet Institute — http://www.bordet.be/